CLINICAL TRIAL: NCT02985073
Title: The Gothenburg TIGR/Veritas® Study - A Comparison Between Biological (Veritas®) vs Non Biological Mesh (TIGR®) in Immediate Breast Reconstruction
Brief Title: A Comparison Between Biological (Veritas®) vs Non Biological Mesh (TIGR®) in Immediate Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 189-16
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Veritas® mesh (Experimental): Use of Veritas mesh in conjunction with immediate breast reconstruction on one side
  Interventions: Device: Veritas®
- TIGR® mesh (Experimental): Use of TIGR® mesh in conjunction with immediate breast reconstruction on one side
  Interventions: Device: TIGR®

INTERVENTIONS:
Device: Veritas® — Biologic mesh
  Arms: Veritas® mesh
Device: TIGR® — Non biologic mesh
  Arms: TIGR® mesh

SUMMARY:
This study compares the outcome using a biological mesh (Veritas®) compared to a non biological mesh (TIGR®) in immediate breast reconstruction.

DETAILED DESCRIPTION:
The scientific evidence using different types of mesh in breast reconstruction is low at present with very few randomized controlled studies.

This study aims to compare a biological mesh (Veritas®) compared to a non biological mesh (TIGR®) in patients with hereditary increased risk of developing breast cancer operated with bilateral immediate breast reconstruction regarding implant loss rate,infections,total complication rate,aesthetic outcome, HQOL (health related quality of Life) and economics.

The patients will be enrolled to the study and sign an informed consent. At the operating theater the patient is randomized either to be reconstructed with Veritas® in one breast and TIGR® in the other breast..

The patients will be followed up according to a specified schedule until one year postoperatively as above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed breast cancer gene mutation or a calculated increased risk > 20% of developing a breast cancer during her lifetime.

Exclusion Criteria:

* All patients that don't fulfill criteria above
* Previous breast surgery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2020-01 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Total complication rate | 12 months
  Total complication rate within one year from surgery

SECONDARY OUTCOMES:
Total infection rate | 30 days
  Total infection rate within 30 days from surgery
Total implant loss rate | 12 months
  Total implant loss rate within one year from surgery
Aesthetic outcome | 12 months
  Aesthetic outcome at one year followup will be assessed by analysis of 3-dimensional pre- and post-op pictures in combination with a panel evaluating different aesthetical units of the breast
HQOL | 12 months
  Three validated questionaries will be used to assess HQOL: EQ-5D,HAD30 and BreastQ. The patient fills in these preoperatively and one year postop

OTHER OUTCOMES:
Cost evaluation | 12 months
  Cost evaluation at one year followup will be evaluated in cooperation with hospital Economists,calculating the total post per patient with or without a mesh.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Kölby, Principal Investigator — Dept of plastic surgery Sahlgrenska University Hospital Gothenburg Sweden
Locations (1):
- Dept . of plastic surgery, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hansson E, Burian P, Hallberg H. Comparison of inflammatory response and synovial metaplasia in immediate breast reconstruction with a synthetic and a biological mesh: a randomized controlled clinical trial. J Plast Surg Hand Surg. 2020 Jun;54(3):131-136. doi: 10.1080/2000656X.2019.1704766. Epub 2019 Dec 20. PMID 31859575
- [Result] Hansson E, Edvinsson AC, Hallberg H. Drain secretion and seroma formation after immediate breast reconstruction with a biological and a synthetic mesh, respectively: A randomized controlled study. Breast J. 2020 Sep;26(9):1756-1759. doi: 10.1111/tbj.13921. Epub 2020 Jun 9. PMID 32515840
- [Result] Hansson E, Edvinsson AC, Elander A, Kolby L, Hallberg H. First-year complications after immediate breast reconstruction with a biological and a synthetic mesh in the same patient: A randomized controlled study. J Surg Oncol. 2021 Jan;123(1):80-88. doi: 10.1002/jso.26227. Epub 2020 Oct 13. PMID 33051871
- [Result] Paganini A, Meyer S, Hallberg H, Hansson E. Are patients most satisfied with a synthetic or a biological mesh in dual-plane immediate breast reconstruction after 5 years? A randomized controlled trial comparing the two meshes in the same patient. J Plast Reconstr Aesthet Surg. 2022 Nov;75(11):4133-4143. doi: 10.1016/j.bjps.2022.08.013. Epub 2022 Aug 23. PMID 36154981
- See also: Full text article — https://pubmed.ncbi.nlm.nih.gov/33051871/
- See also: Full text article — https://pubmed.ncbi.nlm.nih.gov/32515840/